CLINICAL TRIAL: NCT03032133
Title: Pain After Total Knee Arthroplasty With Either Regional or Local Pain Katheter
Brief Title: Pain Control After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Mathys Ltd Bettlach (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TKA pain
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Arthroplasty; Total Knee Replacement; Outcome; Results; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regional pain control (Active Comparator): Regional pain catheter
  Interventions: Procedure: Regional pain control
- Local pain control (Experimental): Local intraarticular pain catheter
  Interventions: Procedure: Local pain control

INTERVENTIONS:
Procedure: Regional pain control — Regional pain catheter
  Arms: Regional pain control
Procedure: Local pain control — Local intraarticular pain catheter
  Arms: Local pain control

SUMMARY:
Patients are randomized to receive pain control after Total Knee Arthroplasty with either a regional pain catheter or a local intraarticular pain catheter. Pain, analgetic use and mobility is asessed.

ELIGIBILITY:
Inclusion Criteria:

* Indication to Total Knee Arthroplasty
* Signed informed consent

Exclusion Criteria:

* Chronic pain
* Allergy against local anaesthetics
* Not understanding study or questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 140 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
pain | daily until day 7 after surgery
  Pain on Visual Analog Scale

SECONDARY OUTCOMES:
analgetics | daily until day 7 after surgery
  Use of additional analgetics
Mobility | daily until day 7 after surgery
  grade of mobility
Function | preoperative, 3 month, 1 year
  Knee Society Score
Patient reported outcome | preoperative, 3 month, 1 year
  Oxford Knee Score
Quality of Life | preoperative, 3 month, 1 year
  EQ 5D

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Lützner, MD, Principal Investigator — TU Dresden
Locations (1):
- Universitätsklinikum Carl Gustav Carus, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No